CLINICAL TRIAL: NCT02461017
Title: Endotracheal Tube Audible Leak Test: What is the Accuracy?
Brief Title: Endotracheal Tube Audible Leak Test
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Madhankumar Sathyamoorthy, Assistant Professor, University of Mississippi Medical Center
Other Study IDs: 2015-0164
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Anesthesia Intubation Complication; Mechanical Ventilation Complication
Keywords: intubation; ventilation; airway; airleak
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endotracheal Leak: Assess for Audible Endotracheal Leak; Assess for Endotracheal Leak with direct visualization under rigid bronchoscope
  Interventions: Other: Assess for Audible Endotracheal Leak; Other: Assess for Endotracheal Leak with direct visualization under rigid bronchoscope

INTERVENTIONS:
Other: Assess for Audible Endotracheal Leak — In supine position, the head will be positioned in neutral position. With fresh gas flow at 2-5L/min, and pop off valve in the anesthesia machine closed and pressure in the inspiratory circuit is slowly increased until an audible leak is heard at the mouth. That pressure will be recorded.
Other: Assess for Endotracheal Leak with direct visualization under rigid bronchoscope — In the same patient position, a flexible nasal laryngoscope will be inserted and positioned superior to the laryngeal inlet by the surgeon. With fresh gas flow at 2-5L/min, and pop off valve in the anesthesia machine closed, the pressure in the inspiratory circuit will be increased slowly until a leak around the TT will be visualized by inspecting the supraglottic area for bubbles or air movement around the TT. The peak pressure at which leak is observed physically will be recorded. This is the end of the study.

SUMMARY:
The endotracheal tube (ETT) leak test (LT), or audible leak test is a widely performed assessment to verify appropriate tube size in neonates, infants and children. However, many factors are known to influence the audible leak test. Even though the test is widely performed, the accuracy has not been evaluated.

DETAILED DESCRIPTION:
The endotracheal tube (ETT) leak test (LT), or audible leak when the peak airway pressures reach 15-30 cmH2O, is a commonly performed assessment to confirm that an endotracheal tube size is appropriate for a child in order to minimize the risk of airway injury and adverse events after removal of ETT. Many factors are known to affect the results of the leak test and variation in results among experienced anesthesiologists may be as great as 38%, but the accuracy of the audible leak test by directly observing the presence of a leak around the ETT has not been evaluated. This study will attempt to use direct visualization of the air leak to correlate to and assess the accuracy of the audible air leak test.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 month (post-natal) and 8 years scheduled for ENT surgery requiring general anesthesia with an endotracheal tube.

Exclusion Criteria:

* Known history of subglottic stenosis
* Known history of recurrent croup
* Known history of endolaryngeal or subglottic lesions
* Parents refusal of participation in study

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 1 month (post-natal) and 8 years scheduled for ENT surgery requiring general anesthesia with an endotracheal tube.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Primary Objective Evidence of an audible endotracheal leak and/or direct visualized endotracheal leak | one year.
  Evidence of an audible endotracheal leak and/or direct visualized endotracheal leak using a flexible nasal laryngoscope positioned superior to the laryngeal inlet.

SECONDARY OUTCOMES:
Secondary Objective Evidence suggesting a relationship between the presence of an audible leak and direct visualization for cuffed and uncuffed TT's | one year.
  Evidence suggesting a relationship between the presence of an audible leak and direct visualization for cuffed and uncuffed TT's.

CONTACTS AND LOCATIONS:
Overall Officials: Madhankumar Sathyamoorthy, MBBS, MS, Principal Investigator — Univeristy of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Suominen P, Taivainen T, Tuominen N, Voipio V, Wirtavuori K, Hiller A, Korpela R, Karjalainen T, Meretoja O. Optimally fitted tracheal tubes decrease the probability of postextubation adverse events in children undergoing general anesthesia. Paediatr Anaesth. 2006 Jun;16(6):641-7. doi: 10.1111/j.1460-9592.2005.01832.x. PMID 16719880
- [Background] Finholt DA, Henry DB, Raphaely RC. Factors affecting leak around tracheal tubes in children. Can Anaesth Soc J. 1985 Jul;32(4):326-9. doi: 10.1007/BF03011335. PMID 4027762
- [Background] Schwartz RE, Stayer SA, Pasquariello CA. Tracheal tube leak test--is there inter-observer agreement? Can J Anaesth. 1993 Nov;40(11):1049-52. doi: 10.1007/BF03009476. PMID 8269566